CLINICAL TRIAL: NCT00507312
Title: Assessment of Myocardial Disease in Man Using Novel Non-invasive Diagnostic Tools
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Suspended while we determine if usable data can be collected from this device.
Sponsor: Prof Henry Krum (Other)
Collaborators: HD Medical Group Ltd (Unknown)
Responsible Party: Sponsor-Investigator, Prof Henry Krum, Prof, Monash University
Organization: Monash University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CP-03/06
Record Dates: First submitted 2007-07-25; First posted 2007-07-26 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Cardiovascular Diseases
Keywords: To assess two new diagnostic devices for detecting early Heart Failure.
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Healthy subjects (with no evidence of cardiovascular disease).
  Interventions: Device: HD medical device (ViScope); Device: CSIRO device
- 2 (Experimental): Patients with risk factors for heart failure
  Interventions: Device: HD medical device (ViScope); Device: CSIRO device
- 3 (Experimental): Patients with heart failure
  Interventions: Device: HD medical device (ViScope); Device: CSIRO device

INTERVENTIONS:
Device: HD medical device (ViScope) — Device
Device: CSIRO device — device

SUMMARY:
This study will be testing two devices which are designed to detect cardiovascular disease in patients as early as possible. As there are now many therapies to prevent and treat this condition it is believed that detecting it early will help reduce the burden of the disease and permit more effective treatment.

The two devices the investigators are testing are the ViScope developed by HD Medical and a device developed by CSIRO. Both of these devices are simple, non-invasive and may provide useful information on how well the heart contracts and relaxes as well as valve function of the heart.

The investigators are planning to enroll 100 healthy subjects, 100 participants with risk factors for heart failure and 300 patients with varying types of heart failure.

The data collected from the experimental devices will be compared to the results from standard tests.

Patients will not have any of their therapies altered as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Have provided consent

Risk factor patients also require:

* Hypertension > 2 years
* Diabetes > 2 years
* Known ischemia, TIA, or stroke
* Arrhythmia; or reduced renal function (eGFR<50 ml/min)

Heart Failure patients also require:

* LVEF <40%
* Receiving standard medication for the treatment of symptomatic systolic heart failure with an NYHA Class of II-IV.

Exclusion Criteria:

Health patients (must not have any of the following):

1. Cardiovascular disease
2. Receiving cardiovascular medication
3. Not in normal sinus rhythm (also required for HF patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-10; Primary Completion 2009-01 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To validate the diagnostic ability of the two devices against echo and clinical data as the "gold standard". | Day 1 (study day)
  We will construct received operative characteristic (Roc) curves for sensitivity and specificity of the HD Medical ViScope and the CSIRO back scatter analysis device in detecting heart failure using echocardiogram and clinical data as the "gold standard".

SECONDARY OUTCOMES:
Correlation of the devices with standard tests such as BP, HR and BNP. | Day 1 (study day)
  * Correlation of device values with echocardiogram parameters of systolic and diastolic function.
  * Correlation of device values with BNP levels.
  * Correlation of device values with heart rate variability measurements.
  * Correlation of device values with pulse wave velocity and systemic arterial compliance assessment measures.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Krum, Professor, Principal Investigator — Monash University / Alfred Hospital
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia